CLINICAL TRIAL: NCT03567265
Title: The Prevalence, Incidence and Factors Associated With Intra-abdominal Hypertension Among Patients Admitted in Intensive Care Units in Uganda-a Multi Center Prospective Study
Brief Title: Intra-abdominal Hypertension and Associated Factors Among Patients Admitted in Intensive Care Units in Uganda.
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Doctor, Makerere University
Other Study IDs: MREC 1254; IAH in ug (Other: makerere university)
Record Dates: First submitted 2018-04-26; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Intra-Abdominal Hypertension
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was carried out to determine the prevalence,incidence and factors associated with intra-abdominal hypertension among patients admitted in three intensive care units in Kampala Uganda.

It was a multi-center prospective cohort study carried out in three intensive care units where 126 patients that met the eligibility criteria were included in the study,demographics,of these were recorded and intra-abdominal pressure measured using the intra-vesical technique at 0,24,and 72 hours.data entry was done using epi-data version 3.1.Data analysis is on going.

DETAILED DESCRIPTION:
Research Question:

What is the prevalence, incidence and associated factors of intra-abdominal hypertension among patients admitted in intensive care units in Uganda?

Rationale for research:

Intra-abdominal hypertension (IAH) is defined as intra-abdominal pressure greater than or equal to 12mmHg. In the developed world, it has been found to be common among critically ill patients and associated with high morbidity and mortality. The world society of Abdominal Compartment Syndrome recommends routine screening for IAH of all critically ill patients upon ICU admission.

Several factors have been arguably associated with intra-abdominal hypertension some of which are common among the critically ill patients in our setting. However Intra-abdominal hypertension has not been given due attention in Ugandan critical care units as evidenced by paucity of data concerning its prevalence, low levels of awareness among critical care medical staff, low levels of screening for IAH and limited routine measurement of intra-abdominal pressure among patients admitted in these units.

Intra-abdominal hypertension if undetected results in multi-organ dysfunction, increased length of ICU stay, morbidity, and mortality.

This study therefore seeks to determine the prevalence, incidence and risk factors of intra-abdominal hypertension among the critically ill in Ugandan ICUs so as to create a basis from which protocols to identify, prevent and manage it may be derived.

General objective:

To determine the incidence, prevalence and factors associated with intra-abdominal hypertension among patients admitted in intensive care units in Uganda.

Specific objectives:

To determine the baseline 24 hour and 72 hour prevalence of intra-abdominal hypertension among patients admitted in intensive care units in Uganda.

To determine the 24 hour and 72 hour incidence of intra-abdominal hypertension among patients admitted in intensive care units in Uganda.

To determine factors associated with intra-abdominal hypertension among patients admitted in the intensive care units in Uganda.

METHODS:

Research design: Multi-center prospective cohort study. This design was chosen in order to achieve better representation of patients in intensive care units in Uganda. It s a prospective study because currently there is paucity of data concerning the subject hence a retrospective analysis could not be done. Also follow up of patients is required to assess factors associated with intra-abdominal hypertension.

All patients admitted to the intensive care units will be recruited in the study. Patients' demographics will be recorded at admission. A urinary catheter shall be inserted and intra abdominal pressure measured at admission, 24 hours, and 72 hours. The patients will then be followed up for 28 day mortality.

Study population:

Sample size: 111 Subjects' state of physical health: seriously ill.

Source of participating subjects:

Mulago National Referral intensive care unit Nakasero hospital limited intensive care unit International Hospital Kampala intensive care unit.

Research procedures:

1. All patients admitted in the intensive care units of the study sites during the study period shall be recruited in the study. A waiver of consent shall be obtained
2. All recruited patients shall be reviewed at T0, T24, and T72 hours T0 defined as 0-3 hours post ICU admission, T24 defined as 24 hours post ICU admission, and T72 as 72 hours post ICU admission.
3. During the study period, the principle investigator and /or research assistants using the data collection tool attached will collect data on day of admission, T72 hours and follow up patients for 28 day mortality.
4. Data collected will include: patients 'demographics, referral source, indication for ICU admission, admission vital parameters, mode of ventilation, ventilation period, length of ICU stay, date of death/discharge from the ICU, 24 hour and cumulative fluid balance and intra-abdominal pressure measurements.
5. The patients shall be catherized using a three way Foleys catheter, the urinary bladder drained and 25mls of normal saline instilled in the bladder. The tubing of the collecting bag will be clamped and the catheter connected to a saline manometer. The pressure will then be measured in centimeters of water at the end of expiration. This will be done at T0, T24 and T72 hours.
6. The patients will then be followed up for 28 day ICU mortality, length of stay in the ICU, and duration of ventilation.

Risks/benefits:

Intra-abdominal pressure measurement using the intra-vesical (bladder) technique is a safe and acceptable procedure worldwide and no complications have been noted.

The intensivists in charge of the units will be notified about patients found to have intra-abdominal hypertension and they will decide the management fit for each patient.

Confidentiality assurances:

1. The patients' identification will be by IP numbers and not individual names
2. The data collected will be saved in multiple storage devices and stored in secure places such as drop box.
3. All saved data copies will be updated on a weekly basis and resaved.

Conflict of interest:

The principle investigator has no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to the three intensive care units and were catheterized Patients admitted for more than 24 hours were recruited in the study Patients aged one year and above.

Exclusion Criteria:

* • Patients in which urethral catheterization was not required

  * The patients that were below one year
  * Patients with contraindications to intra-vesical pressure measurement including: pelvic fracture, haematuria, or neurogenic bladder.
  * Pregnant women
  * Patients admitted for less than 24 hours into the ICU

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled critically ill patients admitted in three intensive care units in Kampala Uganda
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal Hypertension | 6 months
  Intra-abdominal pressure was measured using the intra-vesicular technique.Three measurements were done for each patient at time intervals of 0,24 and 72 hours.This was recorded in a questionnaire, the mean and maximum Intra-abdominal pressure were recorded.Intra-abdominal Hypertension was defined according to the Word Society of Abdominal Compartment Syndrome.

SECONDARY OUTCOMES:
To determine 28_ day ICU mortality of patients with intra-abdominal hypertension. | 6 months
  The patients recruited were followed up to discharge or death in the ICU.Mortality was analyzed using survival analysis method.
To determine duration of mechanical ventilation among patients with intra-abdominal hypertension | 6 months
  The duration of mechanical ventilation for the patients recruited in the study was recorded in days and tabulated in form of median and inter-quartile ranges.
To determine the length of ICU stay among patients with intra-abdominal hypertension | 6 months
  The period of stay of the patients recruited in the study was recorded in days on the questionnaire and tabulated in form of median and inter-quartile ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Phiona Nansubuga, MBCHB, Principal Investigator — Makerere University
Locations (1):
- Nansubuga Phiona, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
publication in a peer review journal